CLINICAL TRIAL: NCT02684071
Title: A Phase II Study of Intraventricular Methotrexate With Systemic Topotecan and Cyclophosphamide in Children With Recurrent or Progressive Malignant Brain Tumors
Brief Title: Phase II Study of Intraventricular Methotrexate in Children With Recurrent or Progressive Malignant Brain Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of additional funding; patients (3) no longer receiving intervention.
Sponsor: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Principal Investigator, Ziad Khatib, Director of Neuro-Oncology, Nicklaus Children's Hospital f/k/a Miami Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCH-CNS-1601
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Recurrent Childhood Medulloblastoma; Recurrent Childhood Ependymoma; Childhood Atypical Teratoid/Rhabdoid Tumor; Embryonal Tumor With Abundant Neuropil and True Rosettes; Metastatic Malignant Neoplasm to the Leptomeninges
Keywords: medulloblastoma, ependymoma, AT/RT, embryonal
MeSH Terms: conditions — Medulloblastoma; Familial ependymoma; Rhabdoid Tumor; Neuroectodermal Tumors, Primitive; Meningeal Carcinomatosis; Ependymoma | interventions — Topotecan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra thecal methotrexate (Experimental): IT methotrexate via Ommaya reservoir with concomitant systemic topotecan and cyclophosphamide
  Interventions: Drug: Intra thecal methotrexate; Drug: topotecan; Drug: cyclophosphamide

INTERVENTIONS:
Drug: Intra thecal methotrexate — IT methotrexate via Ommaya reservoir with concomitant systemic topotecan and cyclophosphamide
  Other Names: Intra thecal methotrexate, topotecan and cyclophosphamide
Drug: topotecan — To be administered in conjunction with methotrexate
  Other Names: Intra thecal methotrexate, topotecan and cyclophosphamide
Drug: cyclophosphamide — To be administered in conjunction with methotrexate and topotecan
  Other Names: Intra thecal methotrexate, topotecan and cyclophosphamide

SUMMARY:
The purpose of this research study is to test an experimental treatment method for recurrent or progressive brain tumors in children aged from 0-22 years. The use of methotrexate and chemotherapy (topotecan and cyclophosphamide) is experimental in this study. This means that their use by themselves or together has not been approved by the U.S. Food and Drug Administration for this usage.

DETAILED DESCRIPTION:
The purpose of this research study is to test an experimental treatment method for recurrent or progressive brain tumors in children aged from 0-22 years. The use of methotrexate and chemotherapy (topotecan and cyclophosphamide) is experimental in this study. This means that their use by themselves or together has not been approved by the U.S. Food and Drug Administration for this usage. This study will attempt to determine via serial MRI scans if methotrexate administration into the lateral or fourth ventricle in combination with systemic intravenous topotecan and cyclophosphamide is effective in reducing tumor burden in the brain and spine for patients with recurrent or progressive brain tumors, including medulloblastoma, ependymoma, PNET (Primitive Neuroectodermal Tumor), atypical teratoid/rhabdoid tumor (AT/RT), and other malignant embryonal tumors. In addition, the study will evaluate the toxicity of the above mentioned experimental treatment during a two-year progression-free survival and survival of children with recurrent malignant brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or progressive supratentorial or posterior fossa tumors with measurable disease on imaging studies of the brain and spine or CSF cytology.
* Tumor histology, including: Medulloblastoma , PNET, or other embryonal tumor, Atypical teratoid/rhaboid tumor (AT/RT), and Ependymoma.
* Leptomeningeal dissemination of a previously diagnosed CNS tumor.
* Diagnosis of tumor pathology will be based upon pathology diagnosis from previous surgeries for patients with recurrent tumors.
* Patients must have received prior radiation before current recurrence, unless the patient is less than 36 months old at diagnosis and has progressed after at least one upfront chemotherapy regimen in which case no prior radiation is required.
* Patients must have a life expectancy of at least 12 weeks as indicated by the patient's oncologist and/or neurosurgeon.
* Lansky or Karnofsky Performance status of at least 50.
* Negative pregnancy test.
* Specific organ function requirements for: Central Nervous System, Bone Marrow, renal and liver.

Exclusion Criteria:

* Patients that do not meet the inclusion criteria above.
* Pregnant or lactating female patients.
* Patients currently enrolled in another experimental treatment protocol.
* Patients with documented allergies to any of the chemotherapy agents used in this study.
* Patient/Parent refuses study participation.
* Patient is severely somnolent or comatose.
* Unable or unwilling to commit to return or to follow-up visits.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Tumor response | 6 months
  MRI response

SECONDARY OUTCOMES:
Toxicity of chemotherapy regimen (topotecan and cyclophosphamide) | 6 months
  Laboratory results, MRI, physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Khatib, MD, Principal Investigator — Nicklaus Children's Hospital
Locations (1):
- Nicklaus Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gururangan S, Petros WP, Poussaint TY, Hancock ML, Phillips PC, Friedman HS, Bomgaars L, Blaney SM, Kun LE, Boyett JM. Phase I trial of intrathecal spartaject busulfan in children with neoplastic meningitis: a Pediatric Brain Tumor Consortium Study (PBTC-004). Clin Cancer Res. 2006 Mar 1;12(5):1540-6. doi: 10.1158/1078-0432.CCR-05-2094. PMID 16533779
- [Background] Slavc I, Schuller E, Czech T, Hainfellner JA, Seidl R, Dieckmann K. Intrathecal mafosfamide therapy for pediatric brain tumors with meningeal dissemination. J Neurooncol. 1998 Jun-Jul;38(2-3):213-8. doi: 10.1023/a:1005940405165. PMID 9696374
- [Background] Yoshimura J, Nishiyama K, Mori H, Takahashi H, Fujii Y. Intrathecal chemotherapy for refractory disseminated medulloblastoma. Childs Nerv Syst. 2008 May;24(5):581-5. doi: 10.1007/s00381-007-0538-8. Epub 2007 Dec 5. PMID 18057943
- [Background] Sandberg DI, Solano J, Petito CK, Mian A, Mou C, Koru-Sengul T, Gonzalez-Brito M, Padgett KR, Luqman A, Buitrago JC, Alam F, Wilkerson JR, Crandall KM, Kuluz JW. Safety and pharmacokinetic analysis of methotrexate administered directly into the fourth ventricle in a piglet model. J Neurooncol. 2010 Dec;100(3):397-406. doi: 10.1007/s11060-010-0210-0. Epub 2010 May 4. PMID 20440538
- [Background] Sandberg DI, Crandall KM, Koru-Sengul T, Padgett KR, Landrum J, Babino D, Petito CK, Solano J, Gonzalez-Brito M, Kuluz JW. Pharmacokinetic analysis of etoposide distribution after administration directly into the fourth ventricle in a piglet model. J Neurooncol. 2010 Mar;97(1):25-32. doi: 10.1007/s11060-009-9998-x. Epub 2009 Aug 18. PMID 19688296
- [Result] Sandberg DI, Crandall KM, Petito CK, Padgett KR, Landrum J, Babino D, He D, Solano J, Gonzalez-Brito M, Kuluz JW. Chemotherapy administration directly into the fourth ventricle in a new piglet model. Laboratory Investigation. J Neurosurg Pediatr. 2008 May;1(5):373-80. doi: 10.3171/PED/2008/1/5/373. PMID 18447671
- See also: Nicklaus Children's Hospital Cancer Center — https://www.nicklauschildrens.org/medical-services/cancer-center.aspx